CLINICAL TRIAL: NCT00812513
Title: Phase II Study of Efficacy of Recombinant Human Platelet-derived Growth Factor (R-Pdf/Gbb) in Healing Wounds Caused by Third Degree Thermal and Electrical Burns.
Brief Title: Efficacy of R-Pdf/Gbb in Healing Wounds Caused by Third Degree Thermal and Electrical Burns
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American Scitech International (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Dr. R. Grewal, American Scitech International
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASI-TEBII1208
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Burns; Electric Burns
Keywords: rhPDGF-BB; Platelet derived growth factor; Burns; Thermal burns; Electric burns
MeSH Terms: conditions — Burns; Burns, Electric | interventions — Gels; Genes, sis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: R-Pdf/Gbb 0.01% gel — rhPDGF 0.01% gel is applied to the wound, then covered with dressing once daily for 3 months
  Other Names: Recombinant human platelet-derived growth factor

SUMMARY:
Platelet Derived Growth Factor (PDGF) is a potent mitogen for a wide range of cell types including fibroblasts, smooth muscle and connective tissue. Recombinant human platelet derived growth factor (R-Pdf/Gbb) has biologic activity similar to endogenous platelet derived growth factor (PDGF). Biologic activity of PDGF includes encouraging chemotaxis and proliferation of cells responsible for wound repair and it augments production of granulation tissue.

The growth factor rhPDGF is found effective in patients having diabetic foot ulcer grade III and IV. The nature of wounds in the third degree burns is similar so far as healing process is concerned.

The purpose of this study is to test the hypotheses that the application of R-Pdf/Gbb 0.01% gel on the third degree thermal and electrical burns will heal these wounds within 3 months and there will be improvement in general condition of the patients without any complications.

DETAILED DESCRIPTION:
The R-Pdf/Gbb is recombinant human platelet-derived growth factor. It has been demonstrated that rhPDGF is effective in enhancing wound healing.

OBJECTIVE: The primary objective of the study is to determine the efficacy of R-Pdf/Gbb gel in treating wounds caused by III degree thermal and electrical burns.

HYPOTHESIS 1: That the applications of R-Pdf/Gbb 0.01% gel on III degree thermal and electrical burns will heal these wounds within 3 months.

HYPOTHESIS 2: Subjects, who having III degree thermal and electrical burns with the treatment of R-Pdf/Gbb 0.01% gel, will show improvement in general condition without any complications.

We aim to test these hypotheses by evaluating the clinical outcome in about 120 patients after three months of treatment with R-Pdf/Gbb 0.01% gel applied once daily.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign Informed consent.
* Patients of both genders.
* Patients between ages of 18 to 75 years.
* Patients having third degree wounds caused by thermal and electrical burns.
* Patients not willing to undergo skin grafting.
* Patients with multiple wounds are considered but each burn wound surface area will be less than 1-8 cm2.
* Wounds with adequate perfusion as assessed with the help of laser Doppler flowmeter.

Exclusion Criteria:

* Patient refuses to sign informed consent.
* Burnt wounds severity less/more than III degree (i.e. I, II, IV degree burns).
* Patients having known neoplasm at the site of application.
* Patients with low serum proteins.
* Patients with uncontrolled hyperglycemia.
* Patients who are taking Ibuprofen.
* Patients with known hypersensitivity to parabens.
* All other burns except thermal and electrical burns.
* Neurological or psychiatric pathologies.
* Women who are pregnant or nursing and women of child bearing age, who are not taking contraceptives or not willing to use them for the period of treatment.
* Local or systemic infection
* Conditions that would interfere with wound healing (diabetes, hypertension, inflammatory diseases treated by corticoids)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Complete healing of the third degree burn wound. | 3 months.

SECONDARY OUTCOMES:
Improvement in general condition of the study subjects without any complications. | 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ratna Grewal, MD, Study Chair — American Scitech International- eCRO; Nani E Mansour, MD, Principal Investigator — Saint Barnabas Medical Center, The Burn Center
Locations (1):
- Saint. Barnabas Medical Center, The Burn Center, Livingston, New Jersey, United States